CLINICAL TRIAL: NCT05435040
Title: Evaluation of Proprioceptive Abilities While Wearing an Elastic Orthosis in Patients With Proprioceptive Knee Deficits
Acronym: CAPROG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A00676-37
Record Dates: First submitted 2022-06-14; First posted 2022-06-28 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Proprioceptive Disorders
Keywords: anterior cruciate ligaments rupture; proprioceptive knee brace; rehabilitation
MeSH Terms: conditions — Somatosensory Disorders

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, interventional, open-label, 1-day clinical investigation in a population of patients with proprioceptive knee deficiency. A randomization will be performed in order to know the order of passage of the 2 conditions: with and without wearing a knee brace.
Masking Description: the clinical trial is carried out in open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- self-comparison (Experimental): The patient will be fitted with proprioceptive knee brace and with no knee brace.
  the patient will perform tests (Y Balance Test, test with Weinstein monofilaments, and Joint Position Sense test) and complete visual analog scales with and without the proprioceptive knee brace in a randomized order.
  There is also a satisfaction questionnaire regarding the proprioceptive knee brace to be completed at the end of the study.
  Interventions: Device: proprioceptive knee brace; Device: No knee brace

INTERVENTIONS:
Device: proprioceptive knee brace — the patient will perform the tests with the knee brace
Device: No knee brace — the patient will perform the tests without the knee brace

SUMMARY:
The objective of the study is to compare, with or without wearing an elastic proprioceptive knee brace, the functional proprioceptive capacity of the knee in patients suffering from proprioceptive deficit.

DETAILED DESCRIPTION:
This proprioceptive deficit is found following various traumas or injuries such as Anterior Cruciate Ligament (ACL) rupture, for example.

The use of joint stabilizers (such as knee braces) will allow an increase in sensory input (particularly at the level of cutaneous mechanoreceptors), and improve the biomechanics of the injured joint.

The objective of the study is to compare, with or without wearing an elastic proprioceptive knee brace, the functional proprioceptive capacity of the knee in patients suffering from proprioceptive deficit.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a proprioception deficit of the knee: detection threshold higher than 2.5° on the TTDPM (Threshold to detect passive motion) test
* Patient whose knee measurements are compatible with the sizes of the proprioceptive knee brace
* Patient having signed a free and informed consent form
* Patient affiliated or entitled to a social security plan

Exclusion Criteria:

* Patient with knee pain on walking greater than or equal to 4 out of 10 on a VAS scale.
* Patient in the early phase of acute trauma to the lower limb
* Patient having worn a knee brace in the 48 hours prior to inclusion
* Pregnant women
* Patient presenting one of the contraindications to the use of the knee brace, indicated in the instructions for use
* Patient with a major cognitive impairment incompatible with participation in a clinical trial
* Patient participating in another clinical investigation conducted to establish the conformity of a DM (Medical Device) impacting the judgment criteria
* Vulnerable patient according to article L1121-6 of the public health code, person subject to a judicial protection measure or unable to consent freely

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Comparison of the functional proprioceptive capacity of the knee in patients with proprioceptive deficit with or without wearing an elastic proprioceptive knee brace. | Day 1 (2 times, after condition 1 and after condition 2)
  The functional proprioceptive capacity of the knee is measured via the 3-axis composite score of the Y Balance Test (YBT). This score corresponds to the average of the 3 maximum distances obtained during the YBT test, normalized by leg length.

SECONDARY OUTCOMES:
Evaluation of tactile sensitivity (baresthesia) with or without wearing the knee brace | Day 1 (2 times, after condition 1 and after condition 2)
  Tactile sensitivity (Baresthesia) via the use of Weinstein monofilaments.
Evaluation of the sensitivity to the position of a joint with or without wearing the knee brace | Day 1 (2 times, after condition 1 and after condition 2)
  Sensitivity to the position of a joint by determining the perception of the position of the leg in space via the JPS (Joint Position Sense) test.
Evaluation of the static stability when using or not the knee brace. | Day 1 (2 times, after condition 1 and after condition 2)
  Static stability level is measured by Visual Analogic Scale (VAS) completed by the patient : 0 corresponds to no stability (worst outcome) and 10 to maximum stability (better outcome).
Evaluation of the stability when walking when using or not the knee brace. | Day 1 (2 times, after condition 1 and after condition 2)
  Stability level when walking is measured by Visual Analogic Scale (VAS) completed by the patient : 0 corresponds to no stability (worst outcome) and 10 to maximum stability (better outcome).
Evaluation of the discomfort level when using or not the knee brace. | Day 1 (2 times, after condition 1 and after condition 2)
  Discomfort level when walking is measured by Visual Analogic Scale (VAS) completed by the patient : 0 corresponds to no discomfort (better outcome) and 10 to maximum discomfort (worst outcome).
Evaluation of the fluidity level when using or not the knee brace. | Day 1 (2 times, after condition 1 and after condition 2)
  Fluidity level is measured by Visual Analogic Scale (VAS) completed by the patient : 0 corresponds to no fluidity (worst outcome) and 10 to maximum fluidity (better outcome).
Evaluation of the range of motion ok the knee level when using or not the knee brace. | Day 1 (2 times, after condition 1 and after condition 2)
  Range of motion of the knee level is measured by Visual Analogic Scale (VAS) completed by the patient : 0 corresponds to no range of motion (worst outcome) and 10 to maximum range of motion (better outcome).
Evaluation of patient satisfaction with the use of the knee brace with a specific questionnaire | Day 1
  Patient satisfaction with the use of the knee brace via a specific questionnaire composed of 15 questions.
Evaluation of the patient's tolerance to the use of the knee brace. | Day 1
  Evaluation of the patient's tolerance to the use of the knee brace through the collection of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Roger OULLION, MD, Principal Investigator — Clinique de la Sauvegarde
Locations (1):
- Clinique de la sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riemann BL, Lephart SM. The Sensorimotor System, Part II: The Role of Proprioception in Motor Control and Functional Joint Stability. J Athl Train. 2002 Jan;37(1):80-4. PMID 16558671
- [Background] Johansson H, Sjolander P, Sojka P. Receptors in the knee joint ligaments and their role in the biomechanics of the joint. Crit Rev Biomed Eng. 1991;18(5):341-68. PMID 2036801
- [Background] Wikstrom EA, Tillman MD, Chmielewski TL, Borsa PA. Measurement and evaluation of dynamic joint stability of the knee and ankle after injury. Sports Med. 2006;36(5):393-410. doi: 10.2165/00007256-200636050-00003. PMID 16646628
- [Background] Fremerey RW, Lobenhoffer P, Zeichen J, Skutek M, Bosch U, Tscherne H. Proprioception after rehabilitation and reconstruction in knees with deficiency of the anterior cruciate ligament: a prospective, longitudinal study. J Bone Joint Surg Br. 2000 Aug;82(6):801-6. doi: 10.1302/0301-620x.82b6.10306. PMID 10990300
- [Background] Han J, Waddington G, Adams R, Anson J, Liu Y. Assessing proprioception: A critical review of methods. J Sport Health Sci. 2016 Mar;5(1):80-90. doi: 10.1016/j.jshs.2014.10.004. Epub 2015 Feb 3. PMID 30356896